CLINICAL TRIAL: NCT01867307
Title: An Open-label Mechanistic Study to Examine the Effect of Oral Empagliflozin (25 mg q.d.) on Kinetics of Renal Glucose Reabsorption in Patients With Type 2 Diabetes Mellitus and Healthy Controls
Brief Title: Effect of Empagliflozin Kinetics on Renal Glucose Reabsorption in Patients With Type II Diabetes and Healthy Controls
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1245.66
Record Dates: First submitted 2013-05-21; First posted 2013-06-04 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (2):
- Healthy Controls (Experimental): healthy controls
  Interventions: Drug: BI 10773
- Patients (Experimental): patients with type 2 diabetes mellitus
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin
  Arms: Patients
Drug: BI 10773 — open label
  Arms: Healthy Controls

SUMMARY:
Single center, 14-day, open-label trial to examine the effect of 25 mg q.d. empagliflozin on kinetics of renal glucose reabsorption in patients diagnosed with type 2 diabetes mellitus and healthy controls

ELIGIBILITY:
Inclusion criteria:

1. T2DM patients and healthy controls aged =18 to <70 at Visit 1.
2. Patients diagnosed with T2DM according to the American Diabetes Association criteria prior to informed consent who are drug-naïve
3. T2DM patients on a stable dose of allowed concomitant medications (as determined by investigator) for 30 days prior to entering the study.
4. T2DM patients with HbA1c between >7 and <10.0% (>53 mmol/mol and <86 mmol/mol) at Visit

Exclusion criteria:

1. Patients with type 1 diabetes mellitus.
2. Patients with uncontrolled hyperglycemia with a fasting plasma glucose level greater than 240 mg/dl after an overnight fast.
3. Patients with a history of clinically significant heart disease (New York Heart Classification greater than class 3; more than non-specific ST-T wave changes on the ECG), peripheral vascular disease (history of claudication), or pulmonary disease as determined by investigator.
4. Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Derived] Abdul-Ghani M, Al Jobori H, Daniele G, Adams J, Cersosimo E, Triplitt C, DeFronzo RA. Inhibition of Renal Sodium-Glucose Cotransport With Empagliflozin Lowers Fasting Plasma Glucose and Improves beta-Cell Function in Subjects With Impaired Fasting Glucose. Diabetes. 2017 Sep;66(9):2495-2502. doi: 10.2337/db17-0055. Epub 2017 Jun 13. PMID 28611037
- [Derived] Al-Jobori H, Daniele G, Cersosimo E, Triplitt C, Mehta R, Norton L, DeFronzo RA, Abdul-Ghani M. Empagliflozin and Kinetics of Renal Glucose Transport in Healthy Individuals and Individuals With Type 2 Diabetes. Diabetes. 2017 Jul;66(7):1999-2006. doi: 10.2337/db17-0100. Epub 2017 Apr 20. PMID 28428225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 subjects were enrolled in the trial; 37 subjects were treated with the trial treatment, 2 subjects were not treated with the trial treatment (1 subject from type 2 diabetes mellitus (T2DM) patients arm and 1 subject from the Healthy subjects arm were not treated)
Groups:
- T2DM Patients: Oral administration of empagliflozin (25 mg once daily) in patients with type 2 diabetes mellitus for 14 days
- Healthy Subjects: Oral administration of empagliflozin (25 mg once daily) in healthy subjects for 14 days
Period: Overall Study
Arm/Group | T2DM Patients | Healthy Subjects
Started | 18 (Started are the treated patients) | 19 (Started are the treated patients)
Completed | 15 | 16
Not Completed | 3 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Other Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Population: The treated set (TS) consisted of all subjects and patients who were treated with at least one dose of empagliflozin.
Groups:
- Total: Total of all reporting groups
Arm/Group | T2DM Patients | Healthy Subjects | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (5.5) | 56.7 (6.3) | 55.9 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Renal Tubular Maximum Reabsorptive Capacity for Glucose (TmG) at End of Empagliflozin Treatment (Day 14)
Description: Change from baseline of renal tubular maximum reabsorptive capacity for glucose (TmG) at end of empagliflozin treatment (Day 14).
  Per-protocol set (PPS): PPS consisted of all subjects and patients in the TS who completed the treatment day 14 clamping study without any relevant deviations either in their treatment regimen or in the performance and timing of the measurements.
Time Frame: Baseline and Day 14
Population: Analysable set (AS): This data set is based on the PPS and excluded all primary endpoint and exploratory endpoint data for one healthy subject due to outlying values that were identified in the subject's TmG and urine splay data.
Measure: Mean (Standard Deviation); unit: (milligram / minute/ 1.73 square meters)
Arm/Group | T2DM Patients | Healthy Subjects
Number analyzed (Participants) | 15 | 15
(milligram / minute/ 1.73 square meters) | -321.7 (214.9) | -256.9 (100.0)
Statistical Analysis 1: Comparison: T2DM Patients; Point estimates of the changes from baseline and 95% Confidence interval around the estimates on treatment day 14 were computed; Test type: Superiority or Other; p < 0.0001, Paired t- test — P-value is from a paired t-test; Median Difference (Final Values) = -220.0, 95% CI 2-sided [-440.6 to -202.7], Standard Error of Mean 55.5 — Difference calculated as (Day 14 - baseline) values
Statistical Analysis 2: Comparison: Healthy Subjects; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value is from a paired t-test; Median Difference (Final Values) = -234.0, 95% CI 2-sided [-312.3 to -201.5], Standard Error of Mean 25.8 — Difference calculated as (Day 14 - baseline) values

ADVERSE EVENTS:
Time Frame: From first drug administration through the residual effect and/or follow-up period, up to 21 days
Arm/Group | T2DM Patients | Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 14/18 | 16/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T2DM Patients (N=18) | Healthy Subjects (N=19)
Genital infection fungal (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Phlebitis (Vascular disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 9 | 6
Micturition urgency (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Pain (General disorders) | 1 | 2
Swelling (General disorders) | 1 | 2
Asthenia (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Infusion site swelling (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Urine output increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.